CLINICAL TRIAL: NCT03308227
Title: Plasma and Lung Tissue Concentrations of Linezolid in Septic Shock Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Southeast University, China (Other)
Collaborators: Cttq (Industry)
Responsible Party: Principal Investigator, Jingyuan,Xu, chief doctor, Southeast University, China
Other Study IDs: 2017ZDSYLL051-P01
Record Dates: First submitted 2017-09-22; First posted 2017-10-12 (Actual); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Septic Shock
Keywords: Linezolid; PK/PD; Septic shock
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental Group: septic shock patients;
- Conrol Group: non-septic shock patients;

SUMMARY:
The study measures the plasma and bronchoalveolar lavage fluid concentrations of linezolid in septic shock patients comparing with non-septic shock patients to confirm the impact of septic shock on PK/PD of linezolid.

DETAILED DESCRIPTION:
A wide array of pathophysiological changes occurring in severe sepsis and septic shock patients may influence antibiotics' pharmacokinetic (PK) properties. The pharmacokinetics and tissue distributions of linezolid achieving effective concentrations are key factors of successful clinical outcomes. To the best of our knowledge, no observational clinical studies are available on the plasma and bronchoalveolar lavage fluid concentrations of linezolid in septic shock patients. Severe pneumonia patients known or suspected to be caused by Gram-positive pathogens will be considered eligible for the study when the attending physician prescribed linezolid as treatment. The plasma and bronchoalveolar lavage fluid concentrations of linezolid are measured in each group at steady state. In an in vitro PK Model, concentration-time curve is drawn to calculate %T>MIC or AUC0-24h/MIC. Linezolid pharmacodynamics evaluation should be based on bacterial eradication and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. between 18 years old and 75 years old;
2. Admitted to the ICU;
3. Expectation, in the opinion of the investigator, that the patients' infection will require ICU stay more than 3 days;
4. Patients diagnosed as severe pneumonia requiring mechanical ventilatory support;
5. Severe pneumonia known or suspected to be caused by Gram-positive pathogens;
6. Expected to treat with linezolid.

Exclusion Criteria:

1. Unable to take bronchoalveolar lavage via bronchofiberscopy;
2. Allergy, hypersensitivity or a serious reaction to linezolid;
3. Treatment with linezolid during the previous 72 hours;
4. Pregnancy.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed as severe pneumonia requiring mechanical ventilatory support.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2017-10-20 (Estimated); Primary Completion 2018-02-28 (Estimated); Study Completion 2018-04-30 (Estimated)

PRIMARY OUTCOMES:
The plasma and bronchoalveolar lavage fluid concentrations of linezolid | Baseline, Day 3, Day 7
  The plasma and bronchoalveolar lavage fluid concentrations of linezolid are measured in each group at steady state

SECONDARY OUTCOMES:
Bacterial eradication | Baseline, Day 3, Day 7
  blood and respiratory secretions culture

OTHER OUTCOMES:
mortality | 28-mortality and 60-mortality
  the outcomes of the patients will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Yingzi Yingzi, PHD, Principal Investigator — Southeast University

IPD SHARING:
Plan to Share IPD: No